CLINICAL TRIAL: NCT06573411
Title: Efficacy and Safety of Finerenone in Patients With Primary Membranous Nephropathy: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Study
Brief Title: Efficacy and Safety of Finerenone in Patients With Primary Membranous Nephropathy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wei Chen, professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIRPRO-PMN
Record Dates: First submitted 2024-08-24; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Primary Membranous Nephropathy
Keywords: finerenone; urinary protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACEI/ARB+finerenone (Experimental): The intervention group will be administered maximum tolerable dose of ACEI/ARB and finerenone 20 mg QD.
  Interventions: Drug: ACEI/ARB+ finerenone
- ACEI/ARB+Placebo (Placebo Comparator): Control patients will be administered maximum tolerable dose of ACEI/ARB and a placebo.
  Interventions: Drug: ACEI/ARB+ Placebo

INTERVENTIONS:
Drug: ACEI/ARB+ finerenone — The intervention group will be administered maximum tolerable dose of ACEI/ARB and finerenone 20 mg QD.
  Arms: ACEI/ARB+finerenone
Drug: ACEI/ARB+ Placebo — Control patients will be administered maximum tolerable dose of ACEI/ARB and a placebo.
  Arms: ACEI/ARB+Placebo

SUMMARY:
This is a prospective, randomized, multicenter, double-blinded, placebo-controlled trial. Eighty-eight patients with primary membranous nephropathy (PMN) will be randomly divided into the intervention and control groups. The intervention group will be administered maximum tolerable dose of ACEI/ARB and finerenone 20 mg QD. Control patients will be administered maximum tolerable dose of ACEI/ARB and a placebo. The primary endpoint is the relative change in urinary protein content from baseline to 6 months.

DETAILED DESCRIPTION:
After more than 4 weeks of maximum tolerated dose of ACEI/ARB, the patients will be randomly divided into the control and intervention groups in a 1:1 ratio in a double-blinded manner. The intervention group will then be administered finerenone 20 mg QD, while control cases will receive a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age≥18,and ≤75) with primary MN.
* Administration of the maximum tolerable dose of ACEI/ARB for ≥4 weeks.
* BP ≤140/90 mmHg.
* Urine protein content of 1.0-5.0 g/d.
* eGFR ≥60 (CKD-EPI).
* Postmenopausal or postoperatively infertile status or on medical contraception (considering the potential risk of thromboembolism in patients with kidney disease) in women.
* Voluntary signing of informed consent.

Exclusion Criteria:

* Type 1 or type 2 diabetes. Patients with a recent history of steroid-induced diabetes were eligible with renal biopsy showing no evidence of secondary diabetic nephropathy within 6 months before the screening period.
* Patients with secondary membranous nephropathy (e.g., due to hepatitis B and C, systemic lupus erythematosus, drug therapy, malignant tumors and other secondary causes).
* Uncontrolled arterial hypertension.
* Treatment with glucocorticoids, immunosuppressants and/or biological agents in the past 6 months.
* Treatment with any other study drug within the last month.
* Females with a positive pregnancy screening test, lactating or planning to become pregnant in the next 24 months. Female or male patients unwilling to use contraceptive methods throughout the study.
* A history of mental illness.
* Laboratory tests meeting the following criteria:

  1. Hemoglobin levels <80 g/L;
  2. Platelet count <80×109/L;
  3. Neutrophil count <1.0×109/L;
  4. Aspartate aminotransferase (AST) or amino aminotransferase (ALT) >2.5 times the upper limit of normal, except in relation to the primary disease.
* Very high-risk cases (life-threatening nephrotic syndrome or unexplained rapid deterioration of renal function).
* Unsuitability for inclusion in the trial as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Relative change in urinary protein content from baseline to 6 months. | 6 months
  To evaluate the effects of ACEI/ARB combined with finerenone on proteinuria in patients with PMN compared to ACEI/ARB alone.

IPD SHARING:
Plan to Share IPD: No